CLINICAL TRIAL: NCT03793127
Title: BAT as a Therapeutic for the Metabolic and Cardiac Dysfunction With Senescence Pilot
Brief Title: Brown Adipose Tissue Pilot
Acronym: BATSP
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMD 1344107
Record Dates: First submitted 2018-12-14; First posted 2019-01-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Aging
MeSH Terms: interventions — glycine N-choloyltransferase; X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young group: 20-40 years of age
  Interventions: Other: Maximal oxygen consumption (V02 max); Other: Brown adipose tissue (BAT) imaging; Other: Muscle function testing
- Old group: 60-80 years of age
  Interventions: Other: Maximal oxygen consumption (V02 max); Other: Brown adipose tissue (BAT) imaging; Other: Muscle function testing

INTERVENTIONS:
Other: Maximal oxygen consumption (V02 max) — Aerobic fitness will be determined by measuring V02 max during a stationary bicycle exercise test.
Other: Brown adipose tissue (BAT) imaging — Brown adipose tissue will be differentiated from white adipose tissue using fat fraction and T2* relaxation time maps generated from a commercially available modified 6-point Dixon (mDixon) water-fat separation method.
Other: Muscle function testing — This test will be done on a machine called a Biodex. We will measure the speed at which subjects move resistance at different percentages of their peak strength.

SUMMARY:
The primary purpose of this protocol is to develop a reliable method to determine BAT mass in young and older adults by magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent and has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.
* Adult female or male, 20-40 or 60-80 years of age, inclusive at time of screening.
* BMI ≥19.0 and ≤34.9 kg/m2, inclusive at time of screening.
* Stable weight (No gain/loss of ≥ 10 lbs within 6 months prior to screening).
* Non-smokers as defined by not smoked any tobacco or nicotine-containing products vape pens or vaporizers within 3 months prior to screening.

Exclusion Criteria:

* History of type 1 or type 2 diabetes per self-report at screening visit 1; or Hgb A1c ≥ 6.5% at screening..
* Actively pursuing weight loss and/or lifestyle changes at time of screening.
* Weight > 450 lbs at screening.
* Uncontrolled hypertension (BP >160 mmHg systolic or >100 mmHg diastolic).
* Mini Mental State Exam (MMSE) <21, only applicable for those 60-80 years of age
* Significant cardiovascular event (e.g. myocardial infarction, stroke) ≤ 6 months prior to screening visit; or stated history of congestive heart failure; or evidence of cardiovascular disease assessed during the ECG at screening.
* Current infection (requiring prescription antimicrobial or antiviral medication, or hospitalization), or corticosteroid treatment (with the exception of inhaled or topical steroids) in the last 3 months prior to screening visit.
* Prescription strength anti-inflammatory medication in the 6 weeks prior to screening.
* Surgery requiring >2 days of hospitalization in the last 3 weeks prior to screening visit.
* Active malignancy or autoimmune disease.
* History of chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV, per self-report.
* History of uncontrolled severe diarrhea, nausea or vomiting within 3 months of screening.
* Uncontrolled severe (including stage III or above) gastrointestinal absorption-related disorders, within 3 months of screening, such as: obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome, gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, ischemic colitis.
* History of drug or alcohol abuse (> 3 drinks per day) within the last 5 years.
* Pregnant, lactating or is within 6 weeks postpartum prior to the screening visit.
* Metal implants (pace-maker, aneurysm clips) based on Investigator's judgment at screening.
* Unable to participate in MRI assessments due to physical limitations of equipment tolerances (e.g. MRI bore size) based on Investigator's judgment at screening.
* Unable to tolerate MRI imaging or claustrophobia.
* Urine albumin-to-creatinine ratio (UACR) ≥300 mg/g in a single urine specimen (per National Kidney Foundation guideline) at screening.
* Impaired renal function: estimated glomerular filtration rate (eGFR) ≤ 50 ml/min/1.73m2 determined at screening.
* Significantly impaired liver function in the opinion of the study PI (mild asymptomatic fatty liver is acceptable), or hepatic enzyme tests are ≥2.5 times normal limit at time of screening.
* Total cholesterol level is ˃300 mg/dL at screening.
* Participant has inadequately treated hyperthyroidism (thyroid stimulating hormone [TSH] below normal range) or hypothyroidism (TSH>ULN (upper limit normal) to <10U/mL and symptomatic, or TSH >10 U/mL) at time of screening.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females in the age ranges 20-40 and 60-80 years were recruited. Potential participants were medically screened to determine good health, weight stable (no gain/loss of ≥ 10 lbs in 6 months prior to screening), and without any contraindication to exercise. Approximately equal numbers of men and women will be recruited. Neither race nor ethnicity were exclusions.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Collection of imaging of BAT by magnetic resonance imaging from 10 participants in each of young and old study groups. | 30 minutes
  Brown adipose tissue will be differentiated from white adipose tissue using fat fraction and T2* relaxation time maps generated from a commercially available modified 6-point Dixon (mDixon) water-fat separation method. The participant may be removed from the magnet and repositioned during the exam in order to determine the same day variability of this method.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coen, PhD, Principal Investigator — Study principal investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodama S, Saito K, Tanaka S, Maki M, Yachi Y, Asumi M, Sugawara A, Totsuka K, Shimano H, Ohashi Y, Yamada N, Sone H. Cardiorespiratory fitness as a quantitative predictor of all-cause mortality and cardiovascular events in healthy men and women: a meta-analysis. JAMA. 2009 May 20;301(19):2024-35. doi: 10.1001/jama.2009.681. PMID 19454641
- [Background] Costantino S, Paneni F, Cosentino F. Ageing, metabolism and cardiovascular disease. J Physiol. 2016 Apr 15;594(8):2061-73. doi: 10.1113/JP270538. Epub 2015 Oct 22. PMID 26391109
- [Background] Kalyani RR, Egan JM. Diabetes and altered glucose metabolism with aging. Endocrinol Metab Clin North Am. 2013 Jun;42(2):333-47. doi: 10.1016/j.ecl.2013.02.010. Epub 2013 Mar 22. PMID 23702405
- [Background] Cypess AM, Lehman S, Williams G, Tal I, Rodman D, Goldfine AB, Kuo FC, Palmer EL, Tseng YH, Doria A, Kolodny GM, Kahn CR. Identification and importance of brown adipose tissue in adult humans. N Engl J Med. 2009 Apr 9;360(15):1509-17. doi: 10.1056/NEJMoa0810780. PMID 19357406
- [Background] van Marken Lichtenbelt WD, Vanhommerig JW, Smulders NM, Drossaerts JM, Kemerink GJ, Bouvy ND, Schrauwen P, Teule GJ. Cold-activated brown adipose tissue in healthy men. N Engl J Med. 2009 Apr 9;360(15):1500-8. doi: 10.1056/NEJMoa0808718. PMID 19357405
- [Background] Saito M, Okamatsu-Ogura Y, Matsushita M, Watanabe K, Yoneshiro T, Nio-Kobayashi J, Iwanaga T, Miyagawa M, Kameya T, Nakada K, Kawai Y, Tsujisaki M. High incidence of metabolically active brown adipose tissue in healthy adult humans: effects of cold exposure and adiposity. Diabetes. 2009 Jul;58(7):1526-31. doi: 10.2337/db09-0530. Epub 2009 Apr 28. PMID 19401428
- [Background] Stanford KI, Middelbeek RJ, Townsend KL, An D, Nygaard EB, Hitchcox KM, Markan KR, Nakano K, Hirshman MF, Tseng YH, Goodyear LJ. Brown adipose tissue regulates glucose homeostasis and insulin sensitivity. J Clin Invest. 2013 Jan;123(1):215-23. doi: 10.1172/JCI62308. Epub 2012 Dec 10. PMID 23221344
- [Background] Berbee JF, Boon MR, Khedoe PP, Bartelt A, Schlein C, Worthmann A, Kooijman S, Hoeke G, Mol IM, John C, Jung C, Vazirpanah N, Brouwers LP, Gordts PL, Esko JD, Hiemstra PS, Havekes LM, Scheja L, Heeren J, Rensen PC. Brown fat activation reduces hypercholesterolaemia and protects from atherosclerosis development. Nat Commun. 2015 Mar 10;6:6356. doi: 10.1038/ncomms7356. PMID 25754609
- [Background] Gunawardana SC, Piston DW. Reversal of type 1 diabetes in mice by brown adipose tissue transplant. Diabetes. 2012 Mar;61(3):674-82. doi: 10.2337/db11-0510. Epub 2012 Feb 7. PMID 22315305
- [Background] Thoonen R, Ernande L, Cheng J, Nagasaka Y, Yao V, Miranda-Bezerra A, Chen C, Chao W, Panagia M, Sosnovik DE, Puppala D, Armoundas AA, Hindle A, Bloch KD, Buys ES, Scherrer-Crosbie M. Functional brown adipose tissue limits cardiomyocyte injury and adverse remodeling in catecholamine-induced cardiomyopathy. J Mol Cell Cardiol. 2015 Jul;84:202-11. doi: 10.1016/j.yjmcc.2015.05.002. Epub 2015 May 9. PMID 25968336
- [Background] Stanford KI, Lynes MD, Takahashi H, Baer LA, Arts PJ, May FJ, Lehnig AC, Middelbeek RJW, Richard JJ, So K, Chen EY, Gao F, Narain NR, Distefano G, Shettigar VK, Hirshman MF, Ziolo MT, Kiebish MA, Tseng YH, Coen PM, Goodyear LJ. 12,13-diHOME: An Exercise-Induced Lipokine that Increases Skeletal Muscle Fatty Acid Uptake. Cell Metab. 2018 May 1;27(5):1111-1120.e3. doi: 10.1016/j.cmet.2018.03.020. PMID 29719226
- [Background] Lynes MD, Leiria LO, Lundh M, Bartelt A, Shamsi F, Huang TL, Takahashi H, Hirshman MF, Schlein C, Lee A, Baer LA, May FJ, Gao F, Narain NR, Chen EY, Kiebish MA, Cypess AM, Bluher M, Goodyear LJ, Hotamisligil GS, Stanford KI, Tseng YH. The cold-induced lipokine 12,13-diHOME promotes fatty acid transport into brown adipose tissue. Nat Med. 2017 May;23(5):631-637. doi: 10.1038/nm.4297. Epub 2017 Mar 27. PMID 28346411
- [Background] Rothwell NJ, Stock MJ. Effects of age on diet-induced thermogenesis and brown adipose tissue metabolism in the rat. Int J Obes. 1983;7(6):583-9. PMID 6686217
- [Background] Graja A, Schulz TJ. Mechanisms of aging-related impairment of brown adipocyte development and function. Gerontology. 2015;61(3):211-7. doi: 10.1159/000366557. Epub 2014 Dec 20. PMID 25531079
- [Background] Yazdanyar A, Newman AB. The burden of cardiovascular disease in the elderly: morbidity, mortality, and costs. Clin Geriatr Med. 2009 Nov;25(4):563-77, vii. doi: 10.1016/j.cger.2009.07.007. PMID 19944261
- [Background] Lowell BB, S-Susulic V, Hamann A, Lawitts JA, Himms-Hagen J, Boyer BB, Kozak LP, Flier JS. Development of obesity in transgenic mice after genetic ablation of brown adipose tissue. Nature. 1993 Dec 23-30;366(6457):740-2. doi: 10.1038/366740a0. PMID 8264795
- [Background] Bartelt A, Bruns OT, Reimer R, Hohenberg H, Ittrich H, Peldschus K, Kaul MG, Tromsdorf UI, Weller H, Waurisch C, Eychmuller A, Gordts PL, Rinninger F, Bruegelmann K, Freund B, Nielsen P, Merkel M, Heeren J. Brown adipose tissue activity controls triglyceride clearance. Nat Med. 2011 Feb;17(2):200-5. doi: 10.1038/nm.2297. Epub 2011 Jan 23. PMID 21258337
- [Background] Guerra C, Koza RA, Yamashita H, Walsh K, Kozak LP. Emergence of brown adipocytes in white fat in mice is under genetic control. Effects on body weight and adiposity. J Clin Invest. 1998 Jul 15;102(2):412-20. doi: 10.1172/JCI3155. PMID 9664083
- [Background] Dulloo AG, Miller DS. Energy balance following sympathetic denervation of brown adipose tissue. Can J Physiol Pharmacol. 1984 Feb;62(2):235-40. doi: 10.1139/y84-035. PMID 6713291
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org

DOCUMENTS (1):
  • Informed Consent Form (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03793127/ICF_000.pdf